CLINICAL TRIAL: NCT00986193
Title: Randomized Comparison of Transapical Transcatheter Treatment Versus Conventional Surgery in Patients With Native Aortic Valve Stenosis
Brief Title: Transapical Transcatheter Treatment Versus Conventional Surgery in Patients With Native Aortic Valve Stenosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: By recommendation from the Data and safety monitoring board
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Odense University Hospital (Other); Danish Heart Foundation (Other)
Responsible Party: Principal Investigator, Evald Hoej Christiansen, MD, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Skejby 2008-1
Record Dates: First submitted 2009-09-25; First posted 2009-09-29 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Valve Stenosis; Stent Valve; Biological Aortic Valve Prosthesis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Aortic Valve Surgery (Active Comparator): Insertion of a biological valve
  Interventions: Procedure: Conventional Aortic Valve Surgery
- Transapical Aortic Valve Implantation (Experimental): Transapical implantation of an Edwards SAPIENtm valve
  Interventions: Procedure: Transapical Aortic Valve Implantation

INTERVENTIONS:
Procedure: Transapical Aortic Valve Implantation — Insertion of a stent valve using catheter-based technique through a mini thoracotomy
  Arms: Transapical Aortic Valve Implantation
Procedure: Conventional Aortic Valve Surgery — Operation using heart-lung machine, with insertion of a biological artificial heart valve
  Arms: Conventional Aortic Valve Surgery

SUMMARY:
This study is a randomised comparison of apical stent valve treatment versus conventional valve surgery in patients with severe aortic valve stenosis.

DETAILED DESCRIPTION:
The purpose of the study is to compare the new established apical stent valve treatment with conventional surgical intervention using biological valve prostheses in patients with severe aortic valve stenosis.

The Edwards-SAPIENTM Transcatheter Heart Valve (Edwards Lifesciences, Irvine, CA) will be used in the stent valve group. The Carpentier-Edwards-Perimount Heart Valve (Edwards Lifesciences, Irvine, CA) will be recommended for the conventional surgery group.(Edwards Lifesciences, Irvine, CA).

Heart centres in the Nordic region with experience (>10 cases) in apical stent valve treatment and in conventional surgical treatment of high risk patients with aortic valve stenosis. The study will be initiated at Aarhus University Hospital, Skejby, Denmark.

Study hypothesis:

As compared to conventional aortic valve substitution in patients aged >75 years, apical stent valve treatment reduces the rates of death, cerebrovascular insult (CVI) and need of dialysis for renal failure 1 month after the treatment.

Primary clinical end-point:

Combined end-point consisting of death, CVI and/or renal failure with need for haemodialysis, 1 month after index treatment.

ELIGIBILITY:
Inclusion Criteria:

* Significant aortic valve stenosis (valve area < 1cm2)
* Age > 75 (years Aarhus University Hospital, Skejby)
* Age > 80 years (other participating centres)
* Operable by conventional surgery AND transapical stent valve implantation
* Expected survival > 1 year following successful treatment
* Accept of participation and in follow-up investigations after adequate information
* Informed consent

Exclusion Criteria:

* Coronary artery disease requiring PCI or CABG
* Earlier cardiac surgery
* Myocardial infarction within 24 hours
* Kidney failure requiring any dialysis
* Ongoing infection
* Acute surgery
* Allergy to ASA or Clopidogrel

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-12; Primary Completion 2011-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Death, CVI and/or renal failure requiring any dialysis | 1 month

SECONDARY OUTCOMES:
Echocardiographic results, valve performance | 1 month with subseguent followup

CONTACTS AND LOCATIONS:
Overall Officials: Evald H Christiansen, MD, Principal Investigator — Skejby Hospital, Aarhus, Denmark
Locations (1):
- Aarhus University Hospital, Skejby, Aarhus N, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided